CLINICAL TRIAL: NCT00859456
Title: A Phase II, Open-label, Non-randomized Trial of Sunitinib in Certain Subtypes of Soft Tissue Sarcomas
Brief Title: Sunitinib in Certain Subtypes of Soft Tissue Sarcomas
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed by pharmaceutical sponsor
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAC2308
Record Dates: First submitted 2009-03-09; First posted 2009-03-11 (Estimated); Results first posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Sarcoma, Soft Tissue
MeSH Terms: conditions — Sarcoma | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sunitinib (Experimental): Patients with unresectable or metastatic angiosarcoma, epithelioid sarcoma-like hemangioendothelioma and Kaposi's sarcoma, either receiving Sunitinib as first-line therapy or failure after no more than 2 prior chemotherapy regimens.
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib — Taken daily PO for a 42 day cycle. This cycle is repeated at least twice.
  A small molecule, multi-targeted receptor tyrosine kinase inhibitor that selectively targets and intracellularly blocks the signaling pathways of receptor tyrosine kinase (RTKs).
  Other Names: Sutent; Sunitinib malate; SU011248

SUMMARY:
The purpose of this study is to determine the clinical response rate (complete response and partial response) in patients with metastatic, locally advanced, or locally recurrent vascular soft tissue sarcoma treated with sunitinib.

DETAILED DESCRIPTION:
Soft tissue sarcomas are rare tumors that arise from mesenchymal tissue from anywhere in the body. While surgical intervention can offer a cure for localized soft tissue sarcoma, treatment of unresectable and metastatic disease is particularly challenging. New treatment options are needed for patients with unresectable or metastatic disease if they progress or cannot tolerate conventional chemotherapy. This study will investigate sunitinib - a novel orally-administered multitargeted tyrosine kinase inhibitor with anti-tumor and antiangiogenic activities.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically-proven diagnosis of angiosarcoma, epithelioid sarcoma-like hemangioendothelioma or Kaposi's sarcoma. Both HIV-Related and HIV-Unrelated Kaposi's patients will be included in the trial. Patients with HIV-Related Kaposi's will be required to have a CD4 count >50 cells/µL and Viral Load < 50 copies/ml. They will also need to be willing to take HAART. They can either have stable Kaposi's on HAART for at least 3 months or have progression of their Kaposi's after having been on HAART for at least 10 weeks.
* Not amenable to surgery, radiation, or combined modality treatment with curative intent.
* Evidence of unidimensionally measurable disease by conventional radiographic techniques. In patients with Kaposi's sarcoma, skin lesions at least 10 mm will be considered measurable disease. Bone lesions, ascites, or lymphangitis of skin or lung are not considered measurable.
* No more than 2 prior chemotherapy regimens for metastatic or unresectable disease. Patients may have received prior bevacizumab or other Tyrosine Kinase Inhibitors, excluding sunitinib. Treatment with bevacizumab or other Tyrosine Kinase Inhibitors will not be counted as prior chemotherapy regimens.
* Four weeks since prior chemotherapy, surgery or radiation therapy and resolution of all toxic effects of any prior therapy, surgical procedure or radiation.
* ECOG performance status 0-2.
* Age 18 or greater.

Exclusion Criteria:

* Patients with a "currently active" second malignancy other than non-melanoma skin cancer or carcinoma in situ of the cervix are not to be registered. Patients who are not considered to have a "currently active" malignancy if they have completed therapy and are considered by their physician to be at less than 30% risk of relapse.
* No areas of measurable disease by CT or MRI.
* Any of the following within the 6 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, or cerebrovascular accident. or transient ischemic attack, or pulmonary embolism.
* Ongoing cardiac dysrhythmias, atrial fibrillation or prolongation of the QTc interval to >450 msec for males of > 470 msec for females. Medications that may prolong the QT intervals should be discontinued or switched to another medication prior to starting Sutent unless determined by the investigator to be absolutely necessary.
* Pregnancy or breastfeeding.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with the study participation or study drug administration.
* Major surgery or radiation therapy within 4 weeks of starting the study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-04 (Actual); Primary Completion 2012-11 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert N Taub, MD, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 subject decided to pursue treatment elsewhere prior to receiving study drug after consent.
Groups:
- Sunitinib: Patients with unresectable or metastatic angiosarcoma, epithelioid sarcoma-like hemangioendothelioma and Kaposi's sarcoma, either receiving Sunitinib as first-line therapy or failure after no more than 2 prior chemotherapy regimens.
  Sunitinib: Taken daily PO for a 42 day cycle. This cycle is repeated at least twice.
  A small molecule, multi-targeted receptor tyrosine kinase inhibitor that selectively targets and intracellularly blocks the signaling pathways of receptor tyrosine kinase (RTKs).
Period: Overall Study
Arm/Group | Sunitinib
Started | 9
Completed | 1
Not Completed | 8
Not completed — Adverse Event | 3
Not completed — Progressive disease | 2
Not completed — Non-compliance | 3

BASELINE CHARACTERISTICS:
Population: 10 subjects were consented; however, 1 subject decided to pursue treatment elsewhere prior to receiving study drug after consent.
Arm/Group | Sunitinib
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Stable Disease at First Assessment of Response
Description: CT or MRI to monitor response: CT or MRI to assess tumor measurement based on the RECIST criteria
Time Frame: Up to 84 days
Measure: Number; unit: participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 9
participants | 6

ADVERSE EVENTS:
Arm/Group | Sunitinib
Serious Adverse Events (participants affected / at risk) | 1/9
Other Adverse Events (participants affected / at risk) | 5/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=9)
Acute Myocardial Infarction (Cardiac disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=9)
Fatigue (General disorders) | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2
Mucositis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Night sweats (General disorders) | 1
Upper Respiratory Infection (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes